CLINICAL TRIAL: NCT07377526
Title: Phase 1/2 Study Of IL15-Transduced, TGFBR2 KO, TROP2 CAR- Engineered Cord Blood-Derived NK Cells Administered Intraperitoneally And Intravenously In Combination With Oral Belzutifan For The Management Of Pancreatic Cancer
Brief Title: Phase 1/2 Study TROP2 CAREngineered Cord Blood-Derived NK Cells + Belzutifan In Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1462; NCI-2026-00667 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2026-01-26; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with TROP2 CAR/IL-15 TGFBR2 KO NK cells + Oral Belzutifan (Experimental): Treatment will be administered on an inpatient basis for lymphodepleting therapy, cell infusion and first doses of belzultifan, and on an outpatient basis after patients are dismissed from the hospital and continue self-administering belzultifan at home.
  Interventions: Drug: TGFBR2 KO CAR27/IL-15 NK cells

INTERVENTIONS:
Drug: TGFBR2 KO CAR27/IL-15 NK cells — Given by mouth

SUMMARY:
This is a Phase I/II study evaluating the intraperitoneal delivery of TROP2 CAR/IL-15 TGFBR2 KO NK cells in combination with oral belzutifan (120 mg daily) for patients with recurrent, locally advanced, unresectable and metastatic pancreatic cancer. The primary objectives are to assess safety and determine the recommended Phase II dose (RP2D).

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety of TROP2 CAR/IL-15 TGFBR2 KO NK cell administered intraperitoneally and intravenously in combination with belzutifan at the flat dose of 120 mg orally daily and define the MTD/RP2D of CAR-NK cells.

Primary Endpoints:

Adverse events as scored by CTCAE V5.0 Dose-limiting toxicity as defined in Section 5.4

Secondary Objectives:

To estimate the best objective response rate (ORR) in patients at 12 weeks after infusion.

To estimate progression-free survival and overall survival. To quantify the persistence of infused allogeneic donor CAR-transduced CB-derived NK cells in the peripheral blood and peritoneal cavity in the recipient. To profile and assess the dynamic changes in the peritoneal tumor microenvironment before and after treatment using single-cell transcriptional and immune profiling on peritoneal cells at various time points before and after treatment. To estimate patient-reported symptom burden and quality of life longitudinally through treatment and follow-up. To compare changes in circulating tumor DNA (ctDNA) with response as determined by RECIST v1.1

Secondary Endpoints:

Objective response rates Progression-free survival Overall survival TROP2 CAR/IL-15 TGFBR2 KO NK cell numbers in peripheral blood and peritoneal cavity vs time profile Characterization of lymphocyte populations at various time points PROMIS-19, EQ-5D-5L, and MDASI-OC PRO questionnaire responses Plasma ctDNA concentration at baselines and serial timepoints

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years or older.
2. Subjects must be willing and able to provide informed consent.
3. Subjects with a histologically confirmed diagnosis of pancreatic ductal adenocarcinoma or ampullary-type carcinoma
4. Subjects who have progressive disease after receiving initial treatment with either FOLFIRINOX, or a gemcitabine-based therapy
5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. A female participant is eligible to participate if at least one of the following conditions applies:

   * Not a woman of childbearing potential (WOCBP) as defined in Appendix 1 OR
   * A WOCBP who agrees to follow the contraceptive guidelines in Appendix 1 during the treatment period and for at least 3 months after the last dose of study treatment.
7. Subjects must have measurable disease present as defined by modified RECIST v1.1
8. Subjects must be at least 5 half-lives from the last cytotoxic chemotherapy at the time of starting lymphodepleting chemotherapy.
9. Subjects must be willing to undergo intraperitoneal port placement and scheduled peritoneal fluid and peripheral blood draws.
10. Agree to sign the consent to the long-term follow-up protocol PA17-0843 to fulfill the institutional responsibilities to various regulatory agencies
11. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years, unless the patient presents with an applicable exclusionary factor, which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.

    Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post-vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CAR NK cell administration.
12. Subjects must have adequate organ function as defined in the following table (Table 2). Specimens must be collected within 10 days prior to the start of study treatment.

Table 2: Adequate Organ Function Laboratory Values Systemic Function Test Laboratory Value

Hematologic Absolute neutrophil count (ANC) ≥1500/µL Platelets ≥100,000/µL Hemoglobin ≥8.0 g/dL (transfusion is allowed)a Renal Creatinine OR Creatinine clearance (CrCl) by Cockcroft-Gault

* 1.5 x ULNb

  ≥30 mL/min for participants with creatinine > 1.5 x ULNb Hepatic Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels > 1.5 x ULN AST (SGOT) and ALT (SGPT) ≤2.5 x ULN (≤5 x ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT)
* 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

  1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the last 2 weeks of the screening test. Participants may be on a stable dose of erythropoietin (≥ approximately 3 months).
  2. Serum creatinine and creatinine clearance (CrCl) should be interpreted and calculated per institutional standard.

     Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies

     Exclusion Criteria:
     1. Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 3 months after the last dose of trial treatment.
     2. If a WOCBP has a positive urine pregnancy test within 72 hours prior to the start of treatment that cannot be confirmed as negative, a serum pregnancy test will be required (see Appendix 1).
     3. Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the PI. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
     4. Has received prior radiotherapy within 2 weeks of the start of the study intervention.

        Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to any non-central nervous system (CNS) disease.
     5. Has received a live vaccine within 30 days prior to the first dose of study drug.

        Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
     6. Is currently receiving another investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
     7. Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
     8. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers.
     9. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
     10. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
     11. History of interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
     12. Active infection requiring systemic therapy.
     13. Known history of uncontrolled Human Immunodeficiency Virus (HIV) infection. Patients with HIV infection and an undetectable viral load may participate.
     14. Known history of chronic Hepatitis B or Hepatitis C virus infection.
     15. Known history of active TB (Bacillus Tuberculosis).
     16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
     17. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
     18. Has had an allogenic tissue/solid organ transplant.
     19. Clinically significant cardiovascular disease within 12 months from the first dose of study intervention, including New York Heart Association (NYHA) Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular event, or cardiac arrhythmia associated with hemodynamic instability. Note: medically controlled arrhythmia would be permitted.
     20. Prolongation of QTcF interval to >480 ms
     21. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. Subjects with known deep vein thrombosis/pulmonary embolism who are under appropriate anticoagulation treatment are eligible.
     22. Radiographic evidence of tumor encasement or invasion of a major blood vessel, or intratumoral cavitation.
     23. Active peritonitis or diverticulitis
     24. Medical or surgical history that in the treating physician's opinion would make the subjective not a suitable candidate for intraperitoneal therapy. Examples would include surgically documented extensive intraperitoneal adhesions or large volume ascites.
     25. History of severe hypersensitivity reaction with biologic therapy (e.g. monoclonal antibodies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Maria Morelli, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org